CLINICAL TRIAL: NCT01468727
Title: Effectiveness of Xylitol Wipes on Infants in Reducing Bacterial Transmission and Colonization From Mother to Child
Brief Title: Study on Use of Xylitol-wipes to Prevent Dental Caries
Acronym: WIPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: A110449
Record Dates: First submitted 2011-11-07; First posted 2011-11-09 (Estimated); Last update posted 2011-11-16 (Estimated); Status verified 2011-11

CONDITIONS: Dental Caries
Keywords: dental caries; mutans streptococci; lactobacilli; bacterial transmission; bacterial colonization
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- xylitol wipe (Experimental)
  Interventions: Dietary Supplement: xylitol wipe
- placebo wipe (Placebo Comparator)
  Interventions: Dietary Supplement: placebo wipe

INTERVENTIONS:
Dietary Supplement: xylitol wipe — Parents were instructed to wipe their infants' teeth and gums three times per day with two wipes each time after feeding in addition to their daily tooth brushing.
  Arms: xylitol wipe
Dietary Supplement: placebo wipe — Parents were instructed to wipe their infants' teeth and gums three times per day with two wipes each time after feeding in addition to their daily tooth brushing.
  Arms: placebo wipe

SUMMARY:
Mutans streptococci (MS) and lactobacillus species (LB) are the two groups of infectious cariogenic (caries-causing) bacteria most strongly associated with dental caries (dental decay). Infants acquire cariogenic bacteria from their mothers early in development via saliva. There have been several studies that have demonstrated a significant reduction in dental caries associated with consumption of the food additive known as xylitol in children and adults. Xylitol is a non-toxic 5 carbon polyol, approved as a food additive by the FDA, that tastes like and behaves like sucrose in humans. Xylitol is used as a sugar substitute to reduce dental caries as it is not fermentable by the caries causing bacteria. In addition, an observed positive beneficial side effect of this sugar substitute is that xylitol has been shown to reduce mother to child bacterial transfer when used by the mother. It is commonly recommended to wipe infants' teeth and gums with a soft cloth to reduce the formation of dental bacterial plaque. Recently wipes have been marketed that contain xylitol to provide a safe sweet sensation for the infant during this cleaning procedure. However, no study has been conducted that assesses the biological effect of applying xylitol directly to the teeth and gums of infants. This study will be conducted to test whether xylitol applied by swab directly to the infant's teeth and gums will effectively reduce bacterial transfer from mother to child. Children age up to two years old whose mothers have high cariogenic bacterial counts will be recruited to use xylitol wipes 3-4 times daily in addition to their normal preventive regimen. This will be a randomized double blinded study where the control group will receive placebo wipes (with no xylitol) and the experimental group will receive the xylitol wipes. The mother-child pair MS and LB bacterial counts and caries score of the children will be measured at baseline, 3 months, 6 months and 1 year. We will contact all patients that were recruited into the study to inquire whether they are willing to return for further follow-up visits at 1, 2, 3, and 4 years post-wipe treatment completion. If successful, this study will support the use of a simple caries preventive measure that could be easily and safely implemented in young children. Ten MS isolates and unique LB colonies will be isolated from each saliva samples to study their genetic diversities and virulence factors.

The investigators will also investigate whether specific MS genes relate to ECC prevention effect of daily xylitol-wipe application using genomic sequencing of MS isolated from current study when the active intervention was applied.

ELIGIBILITY:
Inclusion Criteria:

1. mothers presenting with active dental decay or restorations within the past year (high caries risk)
2. mothers who are the primary caregivers for their child
3. healthy children without systemic disease aged 6 months to two years
4. Infants younger than 6 months who have one or more teeth present

Exclusion Criteria:

1. mother or child with systemic disease
2. antibiotics or medications taken within the previous 3 months that may alter oral flora and saliva flow for mother or child
3. children who primarily receive care in a daycare center or by a caregiver other than the mother

Ages: 6 Months to 35 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 88 (Actual)
Dates: Start 2007-01; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
new decayed surfaces | 1 year

SECONDARY OUTCOMES:
salivary levels of Mutans Streptococci | 3 month, 6 month, 1 year
levels of lactobacilli | 3 month, 6 month, and one year

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

REFERENCES:
- [Derived] Zhan L, Cheng J, Chang P, Ngo M, Denbesten PK, Hoover CI, Featherstone JD. Effects of xylitol wipes on cariogenic bacteria and caries in young children. J Dent Res. 2012 Jul;91(7 Suppl):85S-90S. doi: 10.1177/0022034511434354. PMID 22699675